CLINICAL TRIAL: NCT06771076
Title: Assessment of the Effect of a Cosmetic Cream With CBD and Natural Ingredients on the Recurring Chronic Tendon Pain in Triathletes, Runners, Cyclists, and Swimmers: a Randomized, Crossover, Placebo-controlled, Double-blind Trial
Brief Title: Effects of a CBD and Natural Ingredients Cream on the Chronic Pain of Triathletes, Runners, Cyclists, and Swimmers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vic - Central University of Catalonia (Other)
Collaborators: Uriach Consumer Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CBDTRI001
Record Dates: First submitted 2024-12-19; First posted 2025-01-13 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Tendinopathy; Injuries; Chronic Pain; Sports; Physical Activity
Keywords: CBD; Cannabidiol; Triathlon; Chronic injuries; Running; Cycling; Swimming
MeSH Terms: conditions — Tendinopathy; Wounds and Injuries; Chronic Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will have two periods of one month in which they will use different creams, one containing CBD and natural ingredients, while the other will not. The cream not used during the first month will be the used one in the second month. These periods will be separated by a one-week wash-out.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Both creams will have identical containers (a neutral white tube), with the only difference being that they will be tagged with the letter "A" or "B" (without any additional information on any part of the container).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cream with CBD and natural ingredients - Cream without CBD and natural ingredients (Experimental): During the first month participants will use the cream with CBD and natural ingredients, and during the second month, the cream without CBD and natural ingredients.
  Interventions: Other: Cream with CBD and natural ingredients; Other: Cream without CBD and natural ingredients
- Cream without CBD and natural ingredients - Cream with CBD and natural ingredients (Experimental): During the first month participants will use the cream without CBD and natural ingredients, and during the second month, the cream with CBD and natural ingredients.
  Interventions: Other: Cream with CBD and natural ingredients; Other: Cream without CBD and natural ingredients

INTERVENTIONS:
Other: Cream with CBD and natural ingredients — Topical application of the cream with CBD and natural ingredients on the injured areas, twice per day (after waking up, and before going to bed). A crossover with the other intervention will be done in the next/previous month (depending on the arm).
  Other Names: Cream with CBD
Other: Cream without CBD and natural ingredients — Topical application of the cream without CBD and natural ingredients on the injured areas, twice per day (after waking up and before going to bed). A crossover with the other intervention will be done in the next/previous month (depending on the arm).
  Other Names: Cream without CBD

SUMMARY:
There is a high prevalence of chronic pain in our society, which is detrimental at an individual and country level. Cannabidiol (CBD) has been proposed as a promising treatment for chronic pain, although more high-quality studies are needed in this area. On the other hand, triathlon, running, cycling, and swimming are sports modalities that have an increasing professionalism and importance, albeit not exempt from injuries.

The main goal of this study is to assess the effectiveness of a topical treatment for recurrent chronic pain caused by tendinopathies with a cream containing CBD in triathletes, runners, cyclists, and swimmers. Consequently, the research question for this study is the following: Can the CBD cream be effective in treating chronic pain? The investigators hypothesize that the cream will be able to affect the pain, both in the short and the long term.

The study will be interventional, with a crossover, randomized, and double-blinded design. Two groups of participants will be generated, as well as two treatment options (CBD cream, and a similar one without the CBD). The subjects will apply one of the treatments for one month, followed by a wash-out week without any cream application, and another month with the other treatment. During these weeks, different parameters will be controlled via online questionnaires.

The analyzed variables will include the following: Chronic pain, acute pain, wellness, perceived exertion, quality of life, and satisfaction with the treatment. Different statistical tests will be applied to the collected data, comparing their means and correlations to infer the results.

ELIGIBILITY:
Inclusion Criteria:

* Being a federated triathlete, runner, cyclist, or swimmer.
* Being 18-70 years old.
* Having chronic pain (present at least 3 months before the beginning of the study).
* Having a diagnosis of patellar, Achilles, or iliotibial band tendinopathy for the lower extremities, and/or shoulder rotator cuff or biceps brachii tendinopathy for the upper extremities.
* Training any modality of triathlon, running, cycling, or swimming 4-5 days per week with a minimal training volume of 8 hours per week.
* Having at least 1 year of experience training in triathlon, running, cycling, or swimming.
* Providing at least 80% of the needed data for the study.

Exclusion Criteria:

* Pregnant women.
* People allergic to any of the ingredients of the creams used.
* People with skin injuries in the zones in which the cream has to be applied.
* Using any other pain treatments. Those who use them before the study can still participate if they stop their usage 1 week before the beginning of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2025-01-18 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
Chronic effect of the cream | Through the two 1-month intervention periods.
  Assessment of the pain in the affected zone/s. The measurement will be done once per week (Fridays at night). Assessed using the Oslo Sports Trauma Research Center Overuse Injury Questionnaire (metric: answers to the questions of the instrument).
Acute effect of the cream | Through the two 1-month intervention periods.
  Assessment of the pain in the affected zone/s. The measurement will be done twice per day before applying the cream (after waking up and before going to bed). Besides, the first time the creams are used, the questionnaire will be answered after 5, 10, 15, and 30 minutes. Assessed using a Visual Analog Scale (metric: answer to the question of the instrument). This scale is answered by moving a slider through a line until the desired number is reached, ranging from 0 to 10. Higher scores mean more pain (a worse outcome).

SECONDARY OUTCOMES:
Effect of the cream on wellness | Through the two 1-month intervention periods.
  Assessment of the wellness of the participants on competition day. The measurement will be done before applying the cream, after waking up. Assessed using a preexisting questionnaire (metric: answers to the questions of the instrument).
Effect of the cream on the perceived exertion | Through the two 1-month intervention periods.
  Assessment of the perceived exertion of the participants after competing. The measurement will be done during the first 15-20 minutes after the competition. Assessed using a Borg scale (metric: answer to the question of the instrument). This scale is answered with a number ranging from 0 to 10. Higher scores mean more exertion (a worse outcome).
Effect of the cream on the quality of life | After the two 1-month intervention periods.
  Assessment of the quality of life of the participants after the treatment. The measurement will be done during the morning of the day after each treatment period has finished. Assessed using specific questions of the World Health Organization Quality of Life-BREF questionnaire (metric: answers to the questions of the instrument). These questions are answered with a number ranging from 1 to 5. Depending on the question, a lower or a higher score may be a worse outcome.
Treatment assessment | After the two 1-month intervention periods.
  Assessment of the organoleptic characteristics and the satisfaction with the treatment. The measurement will be done during the morning of the day after each treatment period has finished. Assessed using ad-hoc questionnaires (metric: answers to the questions of the instrument).

CONTACTS AND LOCATIONS:
Overall Officials: Javier Peña López, Ph.D., Principal Investigator — Sport, Exercise, and Human Movement (SEaHM), University of Vic - Central University of Catalonia
Locations (1):
- University of Vic - Central University of Catalonia, Vic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clarsen B, Bahr R, Myklebust G, Andersson SH, Docking SI, Drew M, Finch CF, Fortington LV, Haroy J, Khan KM, Moreau B, Moore IS, Moller M, Nabhan D, Nielsen RO, Pasanen K, Schwellnus M, Soligard T, Verhagen E. Improved reporting of overuse injuries and health problems in sport: an update of the Oslo Sport Trauma Research Center questionnaires. Br J Sports Med. 2020 Apr;54(7):390-396. doi: 10.1136/bjsports-2019-101337. Epub 2020 Feb 14. PMID 32060142
- [Background] Delgado DA, Lambert BS, Boutris N, McCulloch PC, Robbins AB, Moreno MR, Harris JD. Validation of Digital Visual Analog Scale Pain Scoring With a Traditional Paper-based Visual Analog Scale in Adults. J Am Acad Orthop Surg Glob Res Rev. 2018 Mar 23;2(3):e088. doi: 10.5435/JAAOSGlobal-D-17-00088. eCollection 2018 Mar. PMID 30211382
- [Background] McLean BD, Coutts AJ, Kelly V, McGuigan MR, Cormack SJ. Neuromuscular, endocrine, and perceptual fatigue responses during different length between-match microcycles in professional rugby league players. Int J Sports Physiol Perform. 2010 Sep;5(3):367-83. doi: 10.1123/ijspp.5.3.367. PMID 20861526
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712